CLINICAL TRIAL: NCT02941250
Title: Acute Defibrillation Performance of a Novel Can-less Shock Pathway
Acronym: NPC01PRG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NewPace Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC01PRG
Record Dates: First submitted 2016-10-08; First posted 2016-10-21 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2016-10

CONDITIONS: Tachycardia
MeSH Terms: conditions — Tachycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treatment (Experimental): patients receiving ISSD emulator
  Interventions: Device: ISSD emulator

INTERVENTIONS:
Device: ISSD emulator — induced tachy-arrhythmia to be terminated by ISSD emulator

SUMMARY:
Evaluate the operation of the Implantable Subcutaneous String Defibrillator (ISSD) system in patients who require an Implantable Cardioverter Defibrillator (ICD) using an emulator.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the operation, safety, and feasibility of the ISSD system in patients who require an ICD. An ISSD emulator will be briefly implanted and tested during the standard implantation procedure of an ICD, and then entirely removed.

The emulator is not a powered medical device.

This acute intra-operative protocol will test the ability of the ISSD to appropriately convert tachyarrhythmia.

ELIGIBILITY:
Inclusion Criteria:

* Subjects meeting class 1, 2a or 2b indication for ICD implantation
* Age >18
* 32 > Body Mass Index (BMI) > 25
* 190 > Height > 165 cm
* 120 > Waist size > 90 cm

Exclusion Criteria:

* Any condition that precludes the subject's ability to comply with the study requirements, including completion of the study
* Female who is pregnant or breastfeeding;
* Female who is of childbearing age who does not use reliable contraception methods (e.g. contraceptive pills, Intra-Uterine Device, estrogen-containing plasters) or had a positive pregnancy test
* An acute infection requiring antibiotics two weeks prior to surgery
* Participation in any other investigational study in the time ICD implantation is planned, unless there is written consent from the study sponsor;
* Use of the antiarrhythmic drug Amiodarone (Cordarone, Sedacoron, Adenosine or other drugs) in the last 6 months before participation in the clinical trial;
* Existence of large permanent electrodes (e.g. epicardial electrodes), more than 3 permanent endocardial electrodes or any other metal object implanted in the upper part of your body;
* Any of the following cardiac diseases: protracted New York Heart Association (NYHA) class III or IV heart failure , Left Ventricular Ejection Fraction (LVEF) < 20% or an enlarged or hypertrophied heart
* Pulmonary hypertension patient, either with a history of moderate or severe pulmonary hypertension or by estimated pulmonary pressure above 45 (by cardiac echo test).
* Chronic Obstructive Pulmonary Disease (COPD) patient that have been hospitalized in the last 12 months for COPD related reasons, require oxygen support or steroid based therapeutic support.
* Subjects with severely impaired kidney function as measured by a Cockcroft-Gault Glomerular Filtration Rate (GFR) with an estimated GFR ≤ 29.
* Subjects with prior abdominal surgery in the upper abdomen, previous upper abdominal trauma or anatomical deformities of the chest or upper abdomen
* Subjects with known bleeding diathesis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-09; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Defibrillation Threshold (DFT) | immediately following induce tachy-arrhythmia
  lowest shock energy required to terminate tachy-arrhythmia

CONTACTS AND LOCATIONS:
Overall Officials: Petr Neuzil, Prof., Principal Investigator — Chief of Cardiology, Na Homolce Hospital, Prague
Locations (1):
- Nemocnice Na Homolce, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided